CLINICAL TRIAL: NCT04963816
Title: Pediatric Postoperative Analgesia With Quadratus Lumborum Block And Dexamethasone As An Adjuvant In Two Routes With Bupivacaine. Prospective Controlled Clinical Trial
Brief Title: Pediatric Postoperative Analgesia With Quadratus Lumborum Block(QLB) And Dexamethasone As An Adjuvant To Bupivacaine.
Acronym: QLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AHMED ABDELAZIZ SHAMA, Lecturer and consultant of anesthesia and surgical ICU, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34737/6/21
Record Dates: First submitted 2021-06-23; First posted 2021-07-15 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Post Operative Pain; Quadratus Lumborum Block; Pediatric; Abdominal Surgery
Keywords: Quadratus lumborum block in pediatrics; Dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-phosphate; Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A Quadratus Lumborum Block with dexamethasone IV (Active Comparator): QLB with (0.5 mL/kg of bupivacaine 0.25%) and IV dexamethasone (0.1-0.3 mg/kg with a maximum dose 10 mg) added to 5 mL normal saline
  Interventions: Procedure: ultrasound guided quadratus lumborum block; Drug: Dexamethasone Phosphate 4 MG/ML Injectable Solution intravenously; Drug: Bupivacaine Injection
- Group B Quadratus Lumborum Block with dexamethasone locally (Active Comparator): QLB with (0.5 mL/kg of bupivacaine 0.25% plus dexamethasone 0.1 mg/kg), and IV 5 mL normal saline
  Interventions: Procedure: ultrasound guided quadratus lumborum block; Drug: Bupivacaine Injection; Drug: Dexamethasone Phosphate 4 MG/ML Injectable Solution locally
- Group C Quadratus Lumborum Block with bupivacaine alone (Placebo Comparator): Patients will receive QLB (0.5 mL/kg of bupivacaine 0.25%) and IV 5 mL normal saline.
  Interventions: Procedure: ultrasound guided quadratus lumborum block; Drug: Bupivacaine Injection

INTERVENTIONS:
Procedure: ultrasound guided quadratus lumborum block — Ultrasound guided quadratus lumborum block will be done to all groups using curved array transducer 5_2 MHz with the patient in supine position and the block will be done by anterior approach
Drug: Dexamethasone Phosphate 4 MG/ML Injectable Solution intravenously — Using dexamethasone as an adjuvant to bupivacaine in ultrasound guided quadratus lumborum block which will be given intravenously in group A
  Other Names: Dexamethasone as an adjuvant intravenously
  Arms: Group A Quadratus Lumborum Block with dexamethasone IV
Drug: Bupivacaine Injection — Bupivacaine will be given to all groups locally with QLB
  Other Names: Light marcaine
Drug: Dexamethasone Phosphate 4 MG/ML Injectable Solution locally — Using dexamethasone as an adjuvant to bupivacaine in ultrasound guided quadratus lumborum block which will be given locally in Group B
  Other Names: Dexamethasone as an adjuvant locally
  Arms: Group B Quadratus Lumborum Block with dexamethasone locally

SUMMARY:
Studying the post-operative analgesic effect of dexamethasone as an adjuvant to bupivacaine giving intravenously and locally with ultrasound guided quadratus lumborum block(QLB) in pediatrics undergoing abdominal surgeries

DETAILED DESCRIPTION:
After obtaining written informed consent from parents or guardians of all patients, 90 patients (6-12 years old) scheduled for abdominal surgeries operations will be included. Patients will be randomly allocated into three groups, 30 patients in each group. Randomization will be based on computer-generated codes maintained in sequentially numbered opaque envelopes.

Anesthetic Technique:

Anesthesia will be induced with Sevoflurane plus fentanyl (0.5µg/kg) and tracheal intubation will be facilitated with Rocuronium (0.4 mg/kg). Anesthesia will be maintained with Sevoflurane (will be adjusted according to A line autoregressive index (AAI)) and Rocuronium (0.1 mg/kg/dose will be given on the basis of train-of-four neuromuscular monitoring). ECG, noninvasive blood pressure, heart rate, temperature, oxygen saturation, and exhaled CO2 (end tidal CO2) will be continuously monitored during the procedure.

• After induction of anesthesia and before skin incision, a QLB will be performed in all patients in the three groups.

The procedure will be done under ultrasound guidance using curved array transducer 5-2MHz (Sonosite ultrasound system). Echogenic needle, Sono Plex Stim cannula (PAJUNK) 22 gauge and 60 mm length will be used. With the patient in the supine position, the site of the ultrasound and needle entry will be sterilized. The QLB block will be performed by anterior approach. The linear probe will be attached in the area of the triangle of Petit in transverse orientation in lateral abdomen in between the iliac crest and the costal margin, near the posterior axillary line. The muscle planes will be identified until visualizing the quadratus lumborum muscle, at the same plane as the psoas major muscle and the erector spinae. The needle tip is placed at the anterolateral border of the QL at its junction of QL with transversalis fascia outside the anterior layer of the thoracolumbar fascia (TLF) and fascia transversalis, and the local anesthetic will be injected.

Anesthesia will be discontinued when the wound dressing applied, and muscle relaxant will be reversed using (50ug/kg) of neostigmine and atropine (0.02mg/kg) and extubating of the patient will be done. The patient will be transferred to the postoperative care unit (POCU).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients(6-12 years)
* ASA physical status I,II
* Abdominal surgery

Exclusion Criteria:

* Parents refusal or legal guardian's refusal
* Allergy to bupivacaine or dexamethasone
* Contraindications to regional techniques
* Failed QLB
* Infection on site of procedure

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hours
  using the Pediatric Objective Pain Scale (15), where each criterion scores 0 - 2 to give a total score 0 - 10, and a total score of less than 5 mean adequate analgesia.
The duration of analgesia | 24 hours
  the time starting from extubation until analgesia will be required as evidenced by a pain score > 4.

SECONDARY OUTCOMES:
The total amount of paracetamol doses | 24 hours
  paracetamol doses (15 mg/kg per dose) as a rescue analgesic will be needed after the onset of pain
Postoperative vomiting | 12 hours
  vomiting and/or retching without expulsion of gastric content will be recorded by a nurse who will be blinded to study conditions. It will treated if vomiting occurred more than twice in 2 minutes with by granisetron

CONTACTS AND LOCATIONS:
Overall Officials: AHMED A SHAMA, MD, Principal Investigator — Lecturer and consultant of anesthesia and surgical ICU in Tanta University and Faculty of Medicine; SHERIF K ARAFA, MD, Study Chair — ASSISTANT PROFESSOR of anesthesia and surgical ICU; AMIR A EL SAYED, MD, Study Chair — ASSISTANT PROFESSOR of anesthesia and surgical ICU
Locations (1):
- Tanta University, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arafa SK, Elsayed AA, Hagras AM, Shama AAA. Pediatric Postoperative Pain Control With Quadratus Lumborum Block and Dexamethasone in Two Routes With Bupivacaine: A Prospective Randomized Controlled Clinical Trial. Pain Physician. 2022 Oct;25(7):E987-E998. PMID 36288584